CLINICAL TRIAL: NCT04630340
Title: An Innovation Involving Self-Surveillance and Serious Gaming to Increase Smoking Quit Rate: Protocol for a Randomized Controlled Trial
Brief Title: An Innovation to Increase Smoking Quit Rate
Acronym: STEADES-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SingHealth Polyclinics (Other)
Collaborators: Taggle Pte Ltd (Unknown); ITE College West (Unknown)
Responsible Party: Principal Investigator, Tan Ngiap Chuan, Director- Research, SingHealth Polyclinics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/2762
Record Dates: First submitted 2020-09-14; First posted 2020-11-16 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Smoking Cessation
Keywords: carbon monoxide; coach; surveillance; serious games
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Feasibility Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEADES-2 (Intervention) arm (Active Comparator): Subjects in the intervention arm will fill up the questionnaire embedded in the STEADES app and be inducted to the use of STEADES-2 device by the CRC. The CRC will assist to download the STEADES app into the subject's smartphone; demonstrate the use of the app and the procedure for the serious games; and linkage to the virtual coach. The subject will use the STEADES-2 device to assess their smoking status and play the game according to the stipulations in the protocol. The STEADES-2 app provides a portal for the subject to interact with the assigned virtual coach and for motivation messages to be delivered to them. The primary outcome is total smoking cessation as measured by
  1. exhaled breath carbon monoxide using the STEADES-2 device and
  2. urine cotinine level which indicates the nicotine from the cigarette smoking The secondary outcome is the score using the System Usability Scale (SUS) to assess the use and experience in using the STEADES-2 system
  Interventions: Device: STEADES-2
- Usual Care (No Intervention): In the control arm, the subjects will be enrolled into the existing smoking cessation program at the respective polyclinic, which covers smoking cessation advice, together with an exhaled breath analyzed using a commercially available eCO measurement device by a trained nurse counsellor. They will complete a questionnaire and their smoking status will be re-assessed at 12 weeks after their enrolment. The primary outcome is total smoking cessation at the end of the study:
  1. as measured by the exhaled breath carbon monoxide level determined by the STEADES-2 device and
  2. urine cotinine levels which is a marker of nicotine level from smoking

INTERVENTIONS:
Device: STEADES-2 — In this arm, the subjects will use a novel exhaled breath carbon monoxide measurement instrument (STEADES-2) for self surveillance of their smoking status. In addition, the subjects will download the STEADES-2 mobile phone application to pay serious games relating to smoking cessation, receive push-though motivational messages and e-coaching from trained healthcare professionals.
  Arms: STEADES-2 (Intervention) arm

SUMMARY:
An Innovation involving Self-Surveillance and Serious Gaming to Increase Smoking Quit rate: Protocol for a randomized controlled trial.

Abstract Introduction and study aims Smoking is a health hazard associated with cancer, vascular and lung diseases. Current methods to manage smoking cessation have limited success. A recent systematic review suggests increase in smoking cessation potential via serious gaming to attain desirable healthcare outcomes. Outcomes are limited in these studies to demonstrate, quantify, and understand these interventions.

The investigators have demonstrated feasibility of a portable device ("STEADES-1") which allows smokers to measure their exhaled-breath carbon monoxide (eCO) levels, related to their cigarette-smoking intensities. They can relay the eCO measurements via smart-phone applications (app) to their virtual coach to report their smoking cessation progress. The investigators have created an enhanced STEADES-2 system, which incorporates gamification using the eCO data as game element and allows anonymized smokers to compete with each other for the game rewards. It has additional authentication functions and embeds an e-coaching program by trained healthcare professionals.

Methods and analysis This pilot randomized controlled trial aims to evaluate the feasibility and outcomes of the STEADES-2 system in increasing smoking quit rate. The former includes assessing the smokers to monitor their eCO levels; leverage on telesupport via the e-Coaching to raise their motivation; reduce relapse tendencies by playing serious games with fellow smokers. The investigators postulate that the smoking quit rate in smokers in the STEADES-2 intervention group will be higher by 50% than the controls over 12 weeks. This trial will randomly select 20 smokers each into the intervention group and the control group. Smokers in both groups will be compared in terms of complete abstinence from cigarettes as the primary outcome at 12 weeks post-enrolment.

Ethics and dissemination The Institutional Review Board approves the study. The results will be disseminated via conferences and publications.

DETAILED DESCRIPTION:
This overarching aim of this pilot randomized controlled trial is to determine the feasibility of implementing the STEADES system (device and app) in smokers and to compare its effectiveness in increasing their smoking quit rate between the intervention and control groups. Feasibility is demonstrated by quantifying the self-surveillance, serious gaming and engagement of the virtual coaches in the STEADES-2 system. Thus the feasibility is evaluated by the utility rate of the STEADES-2 device by the smokers, transmission rate of the eCO data and frequency of interaction with their virtual coach and gamification rate.

Aims The study aims to determine the proportion of smokers with total abstinence of smoking in the STEADES-2 intervention arm compared to those in the control arm at the end of 12 weeks after study enrolment.

Hypothesis The proportion of smokers with total smoking abstinence in the intervention arm will be 50% higher than those in the control arm at the end of 12 weeks from the time of study recruitment. The total smoking abstinence is defined by both the eCO measurement (0-1pmm) from the STEADES-2 device and the negative result based on the cotinine test kit at 12 weeks.

Method The study is a pilot randomized controlled trial in ambulatory setting at public primary care clinics (polyclinics) in a densely populated, urbanised community in Singapore.

Study sites:

The main site for the implementation of the study will be located at two branches of SingHealth Polyclinics in Pasir Ris and Bedok estates in north-eastern and eastern region of the island state.

Subjects The target subjects are adult smokers aged 21 years and above, who will be recruited at the two sites. Smokers from the other SingHealth Polyclinics can be directed to the study sites by internal referral.

Sample size calculation This is planned as a pilot study to assess the feasibility of this complex intervention involving a multi-component innovation. In addition, the limited funding allows the recruitment of up to 40 smokers, 20 of which will be randomly selected to the intervention arm and another 20 to the control arm.

Randomization Randomization will be carried out centrally at the Research Department office at the institution headquarter. The clinical research coordinator will call in to an administrator to determine the assignment of the consented subject. The administrator will use sealed envelope with a prior sequence of allotment based on random numbers generated by SPSS software to assign the subject to either intervention or controlled arm.

Recruitment process A clinical research coordinator (CRC) will be trained by the investigators on the functions and use of the STEADES-2 system. The CRC will recruit smokers who are referred by the clinical teams at the study sites. They will provide information to the potential subjects using the institution review board's approved study documents which describe the study intent and protocol and address their queries before the subjects endorse the written consent form.

Intervention Subjects in the intervention arm will be inducted to the use of STEADES-2 device by the CRC. The CRC will assist to download the STEADES app into the subject's smartphone; demonstrate the use of the app and the procedure for the serious games; and linkage to the virtual coach.

In the control arm, the subjects will be enrolled into the existing smoking cessation program in the respective polyclinic, which covers smoking cessation advice, together with an exhaled breath analysed using a commercially available eCO measurement device and the STEADES device by a trained nurse counsellor. They will complete a questionnaire and their smoking status will be re-assessed at 12 weeks after their enrolment.

Questionnaire

The questionnaire will collect these data from both groups of subjects:

Demographic characteristics (Year of birth, gender, ethnic group, marital status, highest educational level attained, employment status, estimated annual personal incomes) Smoking Characteristics (Readiness to quit smoking [pre-contemplation, contemplation, preparation, action, maintenance], modified Fagerstrom Test for Nicotine dependence; CAGE questionnaire modified for smoking behaviour; 4 "Cs" Test to assess nicotine addiction [compulsion, control, cutting down, withdrawal symptoms, and consequences]; smoker's profile [stress relief, conditional responses, relief of withdrawal symptoms, elevation of depression mood]; number of cigarettes smoked per day)

Intervention arm only: views and experience with the gamification and the STEADES-2 system; Games Experience Questionnaire (GEQ) and System Usability Scale (SUS) Completion visit The subjects of both arms will make a final study visit at the 12th week post-enrolment. Their smoking status of the subjects will be determined by on-site measurement of the eCO using their STEADES-2 device as well as to detect the presence of nicotine related product using the cotinine test kit. Photo of the STEADES-2 measurement and the cotinine test kit result, together with the study identification number of the subject (excluding identifiable personal data such as facial photo) will be recorded by the CRC to define the outcomes and stored in a secured hard disk for references.

Statistical analysis plan Descriptive statistics will be presented in frequency and percentages. Smoking cessation is defined as both measurements using the STEADES-2 device with results of 0 or 1 ppm and negative cotinine test. Smoking cessation will be assessed with demographics using Chi-square test to identify the profiles of those who quit smoking. Smoking cessation between the intervention and control groups will also be compared using Chi-square test. Cells with less than 5 count will be compared using Fisher's Exact test. Independent t test and Mann Whitney U test will also be used for normally distributed data and non-normally distributed data respectively to compare the difference in scores between the two groups for selected variables.

All analyses will be done using IBM SPSS version 25.0. A p-value of less than 0.05 is considered significant.

An e-library will be embedded in the app for reference to the smokers, including curated video, smoking cessation motivational messages. The resource material includes information on the pharmacies where nicotine replacement products can be purchased, dosing which is compatible with the nicotine dependency of the smokers, tips on cutting down on the number of cigarettes.

Data Repository All activities, device measurement and gameplay on the STEADES App will be uploaded to a centralized server, where it will be displayed for the virtual coaches to monitor. Through their dashboard in the app, the virtual coaches will also be able to communicate and prescribe further activities and advice to the smokers.

Virtual Coaches The clinical team of investigators are multidisciplinary primary care professionals including family physicians, nurses and a pharmacist. They have the training and experience in smoking cessation and will serve as e-coaches to provide advice and support to the smokers. They will be anonymized with the use of a generic term like "coach", who will support the smokers via asynchronous counselling via the app.

Implementation time frame The proposed project will be implemented in phases. Phase 1 (week 1-28) Concurrent development of the STEADES device, app, serious games The development of the STEADES-2 device, app and serious games will be carried out by the technical team members. The clinical team will assemble an e-library of motivational messages and develop an associated algorithm to forward these messages to subjects based on their smoking profiles and trend of eCO data. Scripts will be developed for use by the virtual coaches to interact with the smokers. A training manual for the virtual coaches will be concurrently drafted by the STEADES clinical team.

Phase 2 (week 29-36) The STEADES-2 study protocol will be finalized and submitted to CIRB for ethics approval. Meanwhile, the User Acceptability Testing (UAT) of the STEADES-2 and its integration with the mobile app, serious games, virtual coaching system and the algorithm-based motivational messages will be carried out by both the clinical and technical teams, together with the clinical research coordinator.

Phase 3: (week 37-60) This phase will focus on the implementation of the pilot randomized controlled trial with recruitment to be completed over 12 weeks and follow them up for another 12 weeks.

Phase 4: (week 61-64) The clinical team will audit and analyse the data, interpret the results, share the results via presentations, draft and submit publications to journals.

The study sites at the polyclinics will be test-beds for the STEADES-2 system and programme. If the intervention is proven effective, the integrated system will transform the institution smoking cessation programme and potentially leverage on the research partner in this project to incorporate into local national smoking cessation programme.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who smoke at least one cigarette per day
2. Current user of smartphone which STEADES mobile application can be downloaded
3. Willingness to use the STEADES-2 device to monitor the eCO at least once daily for smoking cessation
4. Willingness to engage the virtual coach at least once weekly during the study period
5. Willingness to play the serious games minimally once daily
6. Ability to provide informed consent and to return the STEADES-2 device to the study team upon completion of the study (for intervention group)

Exclusion Criteria:

1. Non-smoker or ex-smoker who has not smoked any cigarette for the past one month
2. Current user of mobile phone which lacks the function to download mobile application
3. Inability to commit to the study completion or return of the STEADES-2 device at the end of the study (for subjects randomized to the intervention group)
4. Any disability which renders the smoker incapable of providing informed consent independently

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with complete smoking cessation in the intervention and control arms | 12 weeks
  Number of subjects with exhaled carbon monoxide level of 0 ppm and negative cotinine test divided by the total number of the enrolled subjects in each arm x100 (in percentage)
Percentage of subjects with Partial Smoking Cessation in then intervention and control arms | 12 weeks
  Number of subjects with exhaled carbon monoxide level above 1ppm or positive cotinine test divided by the total number of enrolled subjects in each arm x100 (in percentage)
Percentage of subjects who fail Smoking Cessation in the intervention and control arms | 12 weeks
  Number of subjects with exhaled carbon monoxide level above 1ppm and positive cotinine test Divided by the total number of enrolled subjects in each arm x 100 (In percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Ngiap Chuan Tan, Principal Investigator — SingHealth Polyclinics
Locations (1):
- Ngiap Chuan Tan, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jepson RG, Harris FM, Platt S, Tannahill C. The effectiveness of interventions to change six health behaviours: a review of reviews. BMC Public Health. 2010 Sep 8;10:538. doi: 10.1186/1471-2458-10-538. PMID 20825660
- [Background] Movsisyan NK, Varduhi P, Arusyak H, Diana P, Armen M, Frances SA. Smoking behavior, attitudes, and cessation counseling among healthcare professionals in Armenia. BMC Public Health. 2012 Nov 24;12:1028. doi: 10.1186/1471-2458-12-1028. PMID 23176746
- [Background] Abdulateef DS, Ali AJ, Abdulateef DS, Mohesh MI. Smoking Knowledge, Attitude, and Practices Among Health Care Professionals from Sulaymaniyah City/Iraq. Tob Use Insights. 2016 Mar 3;9:1-6. doi: 10.4137/TUI.S38171. eCollection 2016. PMID 26966391
- [Background] Beck RS, Daughtridge R, Sloane PD. Physician-patient communication in the primary care office: a systematic review. J Am Board Fam Pract. 2002 Jan-Feb;15(1):25-38. PMID 11841136
- [Background] Buchhalter AR, Fant RV, Henningfield JE. Novel pharmacological approaches for treating tobacco dependence and withdrawal: current status. Drugs. 2008;68(8):1067-88. doi: 10.2165/00003495-200868080-00005. PMID 18484799
- [Background] Kenny PJ, Markou A. Neurobiology of the nicotine withdrawal syndrome. Pharmacol Biochem Behav. 2001 Dec;70(4):531-49. doi: 10.1016/s0091-3057(01)00651-7. PMID 11796152
- [Background] Daoud N, Jung YE, Sheikh Muhammad A, Weinstein R, Qaadny A, Ghattas F, Khatib M, Grotto I. Facilitators and barriers to smoking cessation among minority men using the behavioral-ecological model and Behavior Change Wheel: A concept mapping study. PLoS One. 2018 Oct 24;13(10):e0204657. doi: 10.1371/journal.pone.0204657. eCollection 2018. PMID 30356254
- [Background] Tan JW, Zary N. Diagnostic Markers of User Experience, Play, and Learning for Digital Serious Games: A Conceptual Framework Study. JMIR Serious Games. 2019 Jul 16;7(3):e14620. doi: 10.2196/14620. PMID 31313660
- [Background] Lu AS, Kharrazi H. A State-of-the-Art Systematic Content Analysis of Games for Health. Games Health J. 2018 Feb;7(1):1-15. doi: 10.1089/g4h.2017.0095. Epub 2018 Jan 2. PMID 29293368
- [Background] Derksen ME, van Strijp S, Kunst AE, Daams JG, Jaspers MWM, Fransen MP. Serious games for smoking prevention and cessation: A systematic review of game elements and game effects. J Am Med Inform Assoc. 2020 May 1;27(5):818-833. doi: 10.1093/jamia/ocaa013. PMID 32330255
- [Result] Xi ZX, Spiller K, Gardner EL. Mechanism-based medication development for the treatment of nicotine dependence. Acta Pharmacol Sin. 2009 Jun;30(6):723-39. doi: 10.1038/aps.2009.46. Epub 2009 May 11. PMID 19434058